CLINICAL TRIAL: NCT00140153
Title: Transdermal Testosterone Gel Prn Application for Hypoactive Sexual Desire Disorder in Women: A Controlled Study
Brief Title: Testosterone in Female Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-3973
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: androgel; female sexuale dysfunction; controlled double-blind; testosterone
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone

INTERVENTIONS:
Drug: testosterone gel (Androgel)

SUMMARY:
The success of sildenafil in the treatment of erectile dysfunction has led to efforts to find similar treatments for prevalent disorders of female sexual dysfunction. Daily transdermal testosterone has been shown to improve sexual function in women after oophorectomy (Shifren et al, Transdermal testosterone treatment in women with impaired sexual function after oophorectomy, New England Journal of Medicine, 343; 682-8, 2000). In laboratory measures of sexual arousal, a single application of transdermal testosterone enhanced vaginal blood and increased erotic fantasy in normal volunteer women in the laboratory setting, four hours after application (Tuiten et al, Can sublingual testosterone increase subjective and physiological measures of laboratory-induced sexual arousal?, Arch Gen Psychiatry, 59;465,2002). We therefore planned a study of transdermal testosterone (25mg) marketed as Androgel in female hypoactive sexual desire disorder. Patients are recruited from the sexology clinics at Soroka Hospital and the Beersheva Mental Health Center. They are randomized to Androgel or placebo and given 10 packets and instructed on application to the abdomen and shoulders, four hours before planned intercourse. Patients unable to discuss planned intercourse with their partner are offered psychosexual counseling and those still unable after three sessions are excluded. After one month patients on active Androgel are crossed over to placebo or vice versa. Patients self-rate sexual response after each intercourse using the Brief Index of Sexual Functioning for Women, and Arizona Sexual Experiences Scale (ASEX)-Female and are rated in interview at the end of each month of treatment using the Sexual Function Questionnaire (SFQ-V1). Our prn technique avoids the androgenizing side effects of continuous daily treatment.

DETAILED DESCRIPTION:
The role of androgens in addition to estrogens in female sexual health has been known for several decades [Davis and Tran 2001]. Recently methods of delivering testosterone other than by injection have made the use of androgens in treatment more available. Testosterone gel is absorbed well [Wang, et al. 2000] and has been shown to be effective in the treatment of hypogonadal men. Doses of 100 mg gel rubbed into skin increased testosterone levels to 30-40 nmoles/L within 8-20 hours. Levels returned to baseline in this study within 1-2 days after cessation of chronic treatment although return to baseline after a single application was not studied.

A recent study [Shifren, et al. 2000] has shown that transdermal continuous patch testosterone dose 150micro g or 300micro g vs. placebo daily during the 12 week study improved sexual health including desire, arousal, and orgasm frequency in women with surgically induced menopause after oophorectomy. Blood levels reached 3.0nmoles/L (5x baseline). Shrifren et al [2000] found no significant side effects with transdermal sustained testosterone treatment. Another study [Goldstat, et al. 2003] looked at transdermal testosterone given in gel, 10mg a day given for 12 weeks in a double-blind design for 31 pre-menopausal women with a mean age of 40 years. The women entered the study presenting with low sexual desire. Testosterone treatment resulted in a significant improvement in psychological general well being and sexual self rating scale. No adverse effects were reported. Blood levels of testosterone increase about 2.5 times baseline to 2.6nmoles/L.

Despite the absence of side effects reported in the small studies for relatively short periods of time done up till now in women with testosterone treatment, in the treatment of a long term disorder such as diminished sexual desire it is reasonable to be concerned with androgenizing side effects. Therefore, it would be extremely useful if testosterone could be given on a prn (as needed) basis before sexual intercourse. Recently Tuiten et al [2000] studied normal volunteer women with vaginal flow measures using photoplethysmography in addition to questionnaire data on sexual arousal after exposure to erotic movies with pre treatment of sublingual testosterone vs. placebo in a single dose sublingually of 0.5mg. Testosterone significantly enhanced vaginal blood flow response to the erotic movies and also the subjective sexual interest, desire and arousal to the movies. The psychophysiological effect was maximal 4 hours after the sublingual testosterone. Blood levels of 25nmol/L testosterone, 10 times baseline, were maximal 10 minutes after sublingual delivery and returned to baseline within 90 minutes.

This study suggested that it may be possible to give transdermal testosterone 4-8 hours before intercourse in couples where the female partner suffers from low sexual interest or desire and /or difficulties in arousal, but where the couple is able to plan intercourse several hours in advance, which is possible in many couples, based on our clinical experience. In such couples androgen could be given on a prn basis and the possibility of side effects with long term use greatly reduced. We therefore propose such a study.

Methods The study will be done as a double-blind randomized crossover study. Women entering the study will be pre-menopausal ages 21-40 with a diagnosis of hypo-active sexual disorder by an experienced sexologist diplomate of the Israel Society for Sexual Therapy. Patients will be accepted for study only if they can plan intercourse with their partner. Patients unable to do so will be offered 3 sessions of counseling about sexual communication and those still unable to plan intercourse after those 3 sessions will be excluded from the study. Patients accepted for the study after written informed consent will be given 8 packets of Testosteron Gel (Androgel) 50mg and shown how to spread the gel on the skin of the lower abdomen or upper shoulders. They will be told that they can use the gel up to twice weekly for one month. Patients will be instructed to spread the gel 4-8 hours before planned intercourse. The patients will be instructed to shower to remove any remaining gel after intercourse. After each intercourse they will fill out the Arizona Sexual Experiences Scale (ASEX)- Female [McGahuey, et al. 2000]. At baseline and at the end of the month they will be interviewed and rated for the month as a whole using the Sexual Function Questionnaire (SFQ-V1) [Quirk, et al. 2002]. They will then be given a package of 8 placebo gels with the same instruction and invited back after a month for another rating. Half of the women will be given placebo and then switched over to active androgen.

We request permission to advertise on the internet and/or in newspapers for symptomatic volunteers for the study.

Possible (but improbable due to the low doses and the prn use) side effects include: Increase in total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol, triglycerides, fasting glucose and insulin; changes in blood counts and changes in liver function tests (serum aspartate aminotransferase, serum glutamyltransferase, serum albumin); hirsutism and acne, increase in facial hair or loss of hair; diarrhea, nipple and breast enlargement or breast pains; headache; elevation of blood pressure, changes in mood or aggressiveness. Slight local skin irritation or dryness of skin. However, as stated before, these side effects are unlikely using prn treatment.

Dose: The recent study of Shifren et al [2000] used continuous transdermal patch and reached blood levels of 3.0nmoles/L (5x baseline) in post-menopausal women, with no side effects over 12 weeks. Goldstat et al [2003] looked at transdermal gel 10mg, which is applied daily but washes off as the day wears on, for 12 weeks with no side effects in pre-menopausal women. They reached blood levels of 2.6nmoles/L (2.5x baseline). Tuiten et al [2000] used sublingual one time dose of 0.5mg, reaching a peak blood level of 25nmoles/L (10x baseline) at 10 minutes which returned to baseline within 90 minutes. We propose to minimize side effects and maximize benefit by single application use of 50mg testosterone in transdermal gel to be used only up to twice a week. Blood levels from this dose from Wang et al [2000] should be about 20nmoles/L. Since patients are instructed to shower after intercourse, these blood levels should exist for only 4-8 hours twice a week. Based on Tuiten et al [2000] a short pulse of testosterone up to these levels is necessary to achieve psychophysiological effects, and thus we request permission to use a dose of 50mg Androgel which would be too high if used daily chronically in women.

ELIGIBILITY:
Inclusion Criteria:

pre-menopausal females, hypoactive sexual disorder, age 21-40, able to plan intercourse with partner -

Exclusion Criteria:

-

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Arizona Sexual Experiences Scale (ASEX)
Sexual Function Questionnaire (SFQ-V1)

CONTACTS AND LOCATIONS:
Overall Officials: RH Belmaker, MD, Study Director — Beersheva Mental Health Center
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel